CLINICAL TRIAL: NCT01649544
Title: Comparison of Treatment of Atrial Fibrillation (AF) Between Surgical Ultrasonic Technology (EPICOR) or Drug Therapy (Cordarone) for Patients With AF Requiring Mitral Valve Surgery
Brief Title: Comparison of Treatment of Atrial Fibrillation (AF) Between Surgical Ultrasonic Technology or Drug Therapy for Patients With AF Requiring Mitral Valve Surgery
Acronym: EPICAF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: End of commercialization of the medical device
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1008058; 2011-A00275-36 (Other: ANSM)
Record Dates: First submitted 2012-07-23; First posted 2012-07-25 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Mitral Valvulopathy; Atrial Fibrillation
Keywords: Mitral valvulopathy; Atrial Fibrillation; Amiodarone; Paroxysmal Atrial Fibrillation; Chronic Atrial Fibrillation; Ultrasound Technique
MeSH Terms: conditions — Heart Valve Diseases; Atrial Fibrillation | interventions — Amiodarone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- EPICOR (Experimental): Cardiac ablation system EPICOR (CE n°0344).
  * ablation device EpicorTM UltraCinchTM LP (Class III device)
  * Positioning system and calibration EpicorTM LP (LP PASTM; device Class IIa)
  * Cable connection EpicorTM LP (unsterile)
  * Ablation Control System EpicorTM LP (Class IIb)
  Interventions: Device: EPICOR
- Amiodarone (Active Comparator): Cordarone :
  400 mg/d during the 2 first months 200 mg/d from 3th to 18th month
  Interventions: Drug: Amiodarone

INTERVENTIONS:
Device: EPICOR — Intraoperatively, in addition to the usual gesture, it will be conducted a systematic exclusion-ligation of the left atrium and the establishment of electrodes atrial and ventricular pacing. The right pulmonary veins are isolated by dissection of the inter-atrial groove and application of the probe by biting on the atrial tissue, the procedure is identical on the left after dissection of the area between the left pulmonary artery and pulmonary veins. The use of ultrasound application will require 10 minutes to around the pulmonary veins using a multi-electrode probe set to deliver an output pulse from 15 to 100 Watts at a frequency from 3.5 to 4.6 MHz. Using EPICOR extends the operating time of 15 minutes.
  Arms: EPICOR
Drug: Amiodarone
  Arms: Amiodarone

SUMMARY:
In pre-operative cardiac surgery, 30 to 40% of patients with mitral valvulopathy have had episodes of paroxysmal atrial fibrillation (PAF) or are in permanent or chronic atrial fibrillation (CAF). According to the 1999 PMSI data, close to 4000 mitral valve interventions were performed in France, in other words, more than 1000 patients present with this condition annually; despite a surgical correction of their valvulopathy, patients presenting with a pre-operative chronic atrial fibrillation remain in fibrillation following surgery despite treatment with anti-arrhythmic agents associated or not with a cardioversion. Thus, the survival rate without AF recurrence is 10% at 1 year and 5% at 2 years in patients with AF prior to surgery; on the other hand, patients in sinus rhythm at the time of surgery and without an antecedent of AF exhibit an incidence of no AF of 90% and 74% at 1 and 2 years, respectively. It has also been shown in numerous studies that the long-term morbidity in patients with atrial valve surgery is higher in those with AF.

For more than 10 years, radio-frequency techniques using the endocavitary approach have shown a greater efficacy in maintaining sinus rhythm than drug therapy even though the techniques are invasive. These radio-frequency techniques were developed and tested during mitral surgery, but, to the investigators knowledge, there is only one randomized study that was carried out in a population with permanent AF using radio-frequency technique via the endocardial approach. Maintenance of sinus rhythm was obtained in only 44.4% of patients versus 4.5% in the control group; these results are not in accordance with the published prospective and retrospective registries using the technique peri-operatively. The principal problem of this study is the absence of medical treatment in the control group. In addition, the use of the radio-frequency technique requires an atriotomy resulting in a prolonged surgical time, which increases the peri-operative morbidity.

Other simpler ablation techniques have been developed, such as the one using ultrasound. In comparison with the radio-frequency method, this latter technique presents numerous advantages including the absence of an atriotomy due to the fact that the epicardial pathway is used, a short procedure time (11 min on average), excellent reproducibility, the transmural character of the lesions, along with the simplicity of application. There is not, to the investigators knowledge, a randomized study comparing the peri-operative ultrasound technique (EPICOR) in mitral valve surgery with the conservative reference treatment, notably mitral valve surgery coupled with long-term amiodarone treatment. In effect, while amiodarone is the most efficacious anti-arrhythmic agent in the long-term, this drug is associated with a high percentage of significant side effects, close to 20% at 2 years. The only available results using the ultrasound technique are the registries pertaining to the follow-up of patients undergoing cardiac mitral or aortic surgery, with an antecedent of AF. The results appear to be encouraging with 85% of cases maintained in sinus rhythm at 12 months in the most recent studies. In this clinical context, a French multi-centric registry evaluated the peri-operative treatment of AF with all of the proposed techniques (cryotherapy, radio-frequency, and ultrasound). The percentage of maintenance of sinus rhythm appears to be lower than in the historical registries, at the level of 60%, but the techniques used in this registry were multiple even if 50% of patients were treated with ultrasound; in addition, there was no randomization and follow-up was only for 6 months.

DETAILED DESCRIPTION:
As a consequence, it is very difficult to have a precise idea, in the literature, of the medium- and long-term efficacy of this technique. Despite a diffusion and utilization of the technique in clinical practice, the efficacy of the ultrasound technique has not been compared, in a standardized manner, with amiodarone, which is the only anti-arrhythmic agent that has shown good efficacy in maintaining post-operative sinus rhythm following cardiac surgery. We propose to undertake an open, prospective, randomized, multicenter study evaluating the efficacy of treatment with ultrasound (EPICOR) in the maintenance of sinus rhythm following mitral surgery in two parallel groups, one group with ablation via ultrasound "EPICOR" and a control group treated with "amiodarone", including a long-term follow-up of 18 months. The strategy in this study necessitates the use of amiodarone in the two groups during the first 2 months followed by a cardioversion in the cases of persistent AF 2 months following surgery in both groups, with a cessation of amiodarone therapy in the ultrasound group and maintenance of therapy in the control group. The parallel treatment with amiodarone in the two groups following the surgical intervention is necessary in order to avoid confounding factors in the analysis. In effect, AF during the postoperative period is frequent and may be considered to be secondary to a number of factors, such as the surgery itself, inflammation, temperature, metabolic disturbances, pericardial effusion, etc. This approach is justified, because if the benefit associated with the peri-operative ultrasound technique is validated, this would allow for a reduction in the use of anti-arrhythmic agents, which are associated with side effects, along with a decrease in long-term morbidity via the resulting maintenance of sinus rhythm. In addition, the technique of ablation via ultrasound could, among others, replace the surgical technique of reference (Cox surgery) for which the principal inconvenience is the prolongation of the time of surgery, resulting in an elevated peri-operative morbidity. Therefore, the principal objective of the study is to compare, at 18 months, the efficacy of surgical treatment with ultrasound (EPICOR) on the maintenance of sinus rhythm following mitral valve surgery in comparison with amiodarone.

ELIGIBILITY:
Inclusion Criteria:

* mitral valvulopathy requiring surgery
* paroxysmal atrial fibrillation or permanent or chronic atrial fibrillation
* Left atrium ≤ 55mm
* consent form signed

Exclusion Criteria:

* thyroid dysfunction
* pregnant
* contraindication of amiodarone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-03; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Atrial Fibrillation episode | At 18 months
  At least one episode of symptomatic AF or asymptomatic sustained [> 10 minutes] documented by an ECG or an R-test changes, occurring between 3 months (after restoration of sinus rhythm by cardioversion if necessary at the end of the 2nd month) and 18th month

SECONDARY OUTCOMES:
Adverse drug effects of Amiodarone | At 18 months
  side effects attributable to treatment with amiodarone and has caused it to stop
major cardiovascular event | At 18 months
  An atrial arrhythmia or heart failure or embolic events
Atrial tachycardia | At 18 months
  Atrial tachycardia whose frequency is between 150 and 250 per minute and shows the appearance of which electrocardiographic waves P positive on D2, D3 and AVF.
Death | At 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Antoine DA COSTA, MD PhD, Principal Investigator — CHU de Saint-Etienne
Locations (5):
- France (5):
  - CHU de Grenoble, Grenoble
  - Hospices Civiles de Lyon, Lyon
  - CHU de Montpellier, Montpellier
  - CHU de Rennes, Rennes
  - CHU de Saint-Etienne, Saint-Etienne